CLINICAL TRIAL: NCT06368791
Title: Evaluation of Easy-to-implement Anti-stress Interventions in a Series of N-of-1 Trials Among Physicians in Residence
Brief Title: Anti-Stress Intervention Among Physicians Study
Acronym: ASIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Valentin Max Vetter, Researcher, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30001479
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Stress, Psychological; Burnout, Psychological; Subjective Stress; Occupational Stress
Keywords: N-of-1 trial; Anti-stress Intervention; Box Breathing; Breathing; Mindfulness
MeSH Terms: conditions — Stress, Psychological; Burnout, Psychological; Subjective Stress; Occupational Stress; Respiratory Aspiration | interventions — Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Box Breathing (Experimental): In the intervention phase of the N-of-1 trial participants are instructed to perform box breathing intervention. During the control phase of the N-of-1 trial, participants are instructed to proceed with their daily activities as usual without engaging in the anti-stress intervention.
  Interventions: Behavioral: Box Breathing; Behavioral: Everyday life control
- Breathing and Mindfulness Exercise (Experimental): In the intervention phase of the N-of-1 trial participants are instructed to perform the guided breathing and mindfulness exercise. During the control phase of the N-of-1 trial, participants are instructed to proceed with their daily activities as usual without engaging in the anti-stress intervention.
  Interventions: Behavioral: Breathing and Mindfulness Exercise; Behavioral: Everyday life control

INTERVENTIONS:
Behavioral: Box Breathing — Participants are guided to find a quite and comfortable spot to sit and unwind. They are then directed to inhale deeply for four seconds, hold that breath for another four seconds, and then exhale slowly over four seconds. Following a brief four-second pause, they begin the next cycle of breathing. To assist with this exercise, participants will have access to a video featuring a red dot tracing a square pattern, moving at the pace needed for the breathing technique.
  Other Names: Tactical Breathing
  Arms: Box Breathing
Behavioral: Breathing and Mindfulness Exercise — The second intervention involves a 10-minute session of guided breathing exercises that blend elements of mindfulness meditation with gentle body movements and controlled breathing. Participants are advised to find a quiet space, sit comfortably, and adopt an upright posture. They are then led through a series of brief exercises, incorporating mild stretches for the upper body and focused, mindful breathing.
  Arms: Breathing and Mindfulness Exercise
Behavioral: Everyday life control — Participants are instructed to not perform the anti-stress intervention and to proceed with their daily activities as usual.

SUMMARY:
Medical practice often comes with high stress. Stress negatively affects our health and well-being and is linked to doctors making mistakes, some of which can be deadly.

In this study, the effect of two quick stress-relief methods on daily stress levels is estimated. The two anti-stress exercises are designed to easily fit into daily routines:

1. Box breathing (6 minutes) is known to reduce stress and lower the heart rate. It is used by the military and law enforcement, among others, to manage stress.
2. Breathing and mindfulness exercise (10 minutes): This guided breathing and mindfulness intervention combines mindful breathing with simple body movements, developed to reduce the perceived level of stress.

The effectiveness of these interventions is being examined in a series of N-of-1 trials. Each participant can choose between the interventions. After being randomly allocated to an individual sequence of one-week intervention and control phases, the study begins. Participants record their stress levels daily over the four-week study period. The intervention is only performed in the intervention phases. Upon completing the study, the stress levels during the intervention phases are compared to those in the control phases. Each participant will receive an individual analysis based on the collected data. In addition, the investigators will estimate the effects at the population level.

Three months after the study, a survey will be sent to the participants to check if the benefits have persisted.

ELIGIBILITY:
Inclusion criteria

* Physicians in training in Germany
* Weekly working time in medical activity of at least 9 hours
* Regular access to a mobile phone on which the "StudyU"-App can be installed
* Informed consent

Exclusion criteria

* Age <18 years
* Specialist training already completed
* No clinical activity during the study period or part of the study period (e.g. vacation, research activity, etc.)
* Participation in another intervention study during the study period
* Does not speak German
* Does yoga more than 4 times a month
* Meditates or performs breathing exercises on average more than 4 days per month
* Confirmed or suspected pregnancy
* Presence of a psychiatric disorder
* Presence of cardiovascular disease
* Presence of respiratory or pulmonary disease
* Presence of a neurological disease
* Substance abuse (for example, alcohol, drugs, or other)
* Planned surgery within the next 6 months
* Doctor's recommendation (or self-assessment) not to perform mindfulness or breathing exercises
* Lack of informed consent
* Employee of the Charité - Universitätsmedizin Berlin (due to data protection reasons, employees of the Charité - Universitätsmedizin Berlin will not be included in this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Daily perceived stress | daily on day 1 to day 28 of the study
  Participants are asked to answer the following question on an analog scale from 1 ("not at all") to 10 ("extremely"): "Overall, how stressful was your day?"
Daily expectation of perceived stress level on the following day | daily on day 1 to day 28 of the study
  Participants are asked to answer the following question on an analog scale from 1 ("not at all") to 10 ("extremely"): "Which level of stress do you expect for the following day?"

SECONDARY OUTCOMES:
Level of agreement between expected and actually perceived level of stress | daily on day 1 to day 28 of the study
  By subtracting the expected from the actually experienced level of stress, the level of agreement will be assessed.
Compliance with the study protocol: number of participant reported outcomes | After 4 weeks
  Compliance with the study protocol will be assessed by counting the number of participant reported outcomes documented.
Compliance with the study protocol: number of performed anti-stress interventions | After 4 weeks
  Compliance with the study protocol will be assessed by counting the number of anti-stress interventions completed over the entire duration of the study.
Successful study completion | After 4 weeks
  Successful completion of the study will be assessed based on the minimum required number of results reported by participants during the study period to be included in the final statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin M Vetter, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT06368791/SAP_000.pdf